CLINICAL TRIAL: NCT01700153
Title: Study of the Effectiveness of an Interactive Robot for the Rehabilitation of the Upper Limb in Children With Cerebral Palsy by Evaluating the 3 Fields of the ICF: A Prospective, Randomized, Controlled, Simple Blind Study.
Brief Title: Efficacy Study of an Interactive Robot for the Rehabilitation of the Upper Limb in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Lejeune, Professor, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IONS-Gilliaux-01
Record Dates: First submitted 2012-09-26; First posted 2012-10-04 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Cerebral Palsy
Keywords: Robotic-assisted therapy; cerebral palsy; ICF
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental: Robotic-assisted therapy (Experimental): All patients will receive a similar classical rehabilitation as a basis. the 10 patients of this group will receive a supplement of robotic-assisted therapy.
  Interventions: Other: Robotic-assisted therapy; Other: Classical therapy
- Classical therapy (Active Comparator): All patients will receive a similar classical rehabilitation as a basis. the 10 patients of this group will receive a supplement of classical rehabilitation.
  Interventions: Other: Classical therapy

INTERVENTIONS:
Other: Robotic-assisted therapy — This robotic device is designed to intensively rehabilitate the upper limb. Indeed, this robot allows the patient to perform a lot of active, passive, or assisted exercises. The level of assistance is determined and provided by the robot in function of the patient capacity.
  Arms: Experimental: Robotic-assisted therapy
Other: Classical therapy — conventional therapy will be performed by therapists specialized in neuro-pediatric rehabilitation

SUMMARY:
Cerebral Palsy (CP) is a major cause of impairments in child population. This disease justifies an intensive and prolonged multidisciplinary rehabilitation which can be optimised by robotics.

Our team has developed a robot designed to rehabilitate the child's upper limb. This robot allows the patient to perform active, passive, or assisted exercises.

This therapy is designed to promote motor development in children with CP. Its finality is to improve patients' quality of life and participation.

Several pilot studies evaluated the efficacy of robotic assisted therapy in children with CP but none RCT has been done.

Then, the aim of the study is to evaluate the efficacy of robotic-assisted therapy in children with cerebral palsy by evaluating the 3 fields of the ICF (International Classification of Functioning, Disability and Health) and performing a prospective randomized controlled single blind trial. Therefore, all patients will benefit from a classical rehabilitation as a basis. Furthermore, patients of the control and experimental groups will receive a supplement of classical rehabilitation and robotic-assisted therapy, respectively.

DETAILED DESCRIPTION:
INTRODUCTION

Cerebral Palsy (CP) is a major cause of impairments in child population. Indeed, CP affects two births per thousand (1). The brain damage is expressed by different neurological impairments and functional disabilities. These disabilities justify intensive and sustained multidisciplinary rehabilitation to reduce neurological impairments, to improve the activities and participation of patients, and, ultimately, their quality of life (2, 3, 4).

Robotics interest has already been shown for lower limb rehabilitation (5). The development of the upper limb rehabilitation robotic devices started later. To better stimulate brain plasticity, these tools meet the actual recommendations existing in CP's rehabilitation (4). Indeed, the robots allow the execution of a large number of movements whose quality is controlled (6). A visual interface gives the patient a feedback of its movements (7), and offers exercises oriented functional tasks that have meaning for him (8) and the possibly dive into a virtual reality. All these elements justify the clinical development of robots to assist the therapists.

In children with CP, several pilot studies have verified the clinical applicability of these tools (9-11). However, no randomized controlled study has been performed to evaluate the effectiveness of robotic-assisted therapy in children with CP (12). Moreover, no study evaluated the effect of these therapies on the three areas of the ICF : Many studies focus on impairments (e.g. muscle) without assessing the functional capacity of the patient: what about their ability in every day life?

OBJECTIVES

To perform a prospective, randomized, controlled, single blind trial to assess the efficacy of robotic-assisted therapy in children with cerebral palsy by evaluating the three fields of the ICF.

METHODS

Twenty patients enrolled at the "Institut Royal de l'Accueil du Handicap Moteur" (IRAHM) (1200 Brussels) will be included according to the following criteria: CP, whose location is unilateral (hemiplegia) or bilateral (diplegia, quadriplegia), with a MACS (Manual Ability Classification System) score > 1 (moderate to severe motor impairments) (13). The exclusion criteria are the following: injection in the upper member of botulinum toxin within 6 months or intrathecal baclofen used for the upper limb, an unstable clinical condition contraindicating the upper limb rehabilitation treatments, cognitive disorders preventing the understanding of the instructions or other neurological or orthopedic pathology affecting the upper limb.

A randomisation of patients in two groups (control and experimental) will be performed, using a stratified randomization method to ensure the equivalence of the two groups for age, the location of the symptoms (diplegia, quadriplegia, left or right hemiplegia) and motor neurological impairments (MACS score).

At IRAHM, each child benefits of 3 physiotherapy sessions and 2 occupational therapy sessions per week. Each session lasts 45 minutes. The children in the control group will see no change in their treatment. In the experimental group, 1 physiotherapy session and 1 occupational therapy session will be replaced by two sessions of intensive rehabilitation of the arm with the robot. In total for each group, each child will benefit from 40 sessions of 45 minutes over 8 weeks therapy

Patients will be evaluated three times in the study: before the start of treatments, at the end of treatments, and 3 months after the end of treatments.

Functional assessments will be carried out according to a protocol exploring the three fields of the ICF. Impairments will be evaluated by the score of Quality of Upper Extremity Skills Test (14), MACS (13), and the Box and Block test (15). Then, spasticity (with two scales), kinematics and strength of the paretic arm will be evaluated using the modified Ashworth and Tardieu scales, the ReaPLAN robot and a dynamometer, respectively (9, 16, 17). Disability will be evaluated via Abilhand-kids (18) and Pediatric Evaluation of Disability Inventory (19). Participation restrictions will be evaluated via the MHAVIE questionnaire (20). All assessments will be carried out by a occupational therapist, which will be not informed the group that the child is assigned (single-blind). All rehabilitation and assessment sessions will be conducted at the IRAHM.

PERSPECTIVES

From this study, we hope to demonstrate the efficacy of robotic-assisted therapy in children with cerebral palsy by evaluating the three fields of the ICF. These results could prove that this tool can be a significant complement for the CP rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy (hemi, quadri or di-plegia)
* MACS > 1/5 (moderate to severe impairments)

Exclusion Criteria:

* Botulinum toxin injection in the upper limb muscles
* Intrathecal Baclofen for the upper limb spasticity
* an unstable clinical condition contraindicating the upper limb rehabilitation treatments
* cognitive disorders preventing the understanding of the instructions
* other neurological or orthopedic pathology affecting the upper limb.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Kinematic | Change from Baseline in Kinematic at an expected average of 3 months and 6 months

SECONDARY OUTCOMES:
Manual Ability Classification System | Change from Baseline in manual ability at an expected average of 3 months and 6 months
Quality of Upper Extremity Skills Test | Change from Baseline in quality of upper extremity skills at an expected average of 3 months and 6 months
Box and Block test | Change from Baseline in dexterity at an expected average of 3 months and 6 months
strength | Change from Baseline in strength at an expected average of 3 months and 6 months
Abilhand-Kids scale | Change from Baseline in activity of daily living at an expected average of 3 months and 6 months
Pediatric Evaluation of Disability Inventory | Change from Baseline in activity of daily living at an expected average of 3 months and 6 months
MHAVIE | Change from Baseline in parents' satisfaction of children activity daily living at an expected average of 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Gilliaux, PhD student, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Institut royal de l'accueil du handicap moteur, Brussels, Belgium

REFERENCES:
- [Background] Bax MC, Flodmark O, Tydeman C. Definition and classification of cerebral palsy. From syndrome toward disease. Dev Med Child Neurol Suppl. 2007 Feb;109:39-41. No abstract available. PMID 17370481
- [Background] Duncan PW, Zorowitz R, Bates B, Choi JY, Glasberg JJ, Graham GD, Katz RC, Lamberty K, Reker D. Management of Adult Stroke Rehabilitation Care: a clinical practice guideline. Stroke. 2005 Sep;36(9):e100-43. doi: 10.1161/01.STR.0000180861.54180.FF. No abstract available. PMID 16120836
- [Background] Ward NS. The neural substrates of motor recovery after focal damage to the central nervous system. Arch Phys Med Rehabil. 2006 Dec;87(12 Suppl 2):S30-5. doi: 10.1016/j.apmr.2006.08.334. PMID 17140877
- [Background] Aisen ML, Kerkovich D, Mast J, Mulroy S, Wren TA, Kay RM, Rethlefsen SA. Cerebral palsy: clinical care and neurological rehabilitation. Lancet Neurol. 2011 Sep;10(9):844-52. doi: 10.1016/S1474-4422(11)70176-4. PMID 21849165
- [Background] Mehrholz J, Werner C, Kugler J, Pohl M. Electromechanical-assisted training for walking after stroke. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD006185. doi: 10.1002/14651858.CD006185.pub2. PMID 17943893
- [Background] Masiero S, Celia A, Rosati G, Armani M. Robotic-assisted rehabilitation of the upper limb after acute stroke. Arch Phys Med Rehabil. 2007 Feb;88(2):142-9. doi: 10.1016/j.apmr.2006.10.032. PMID 17270510
- [Background] Housman SJ, Scott KM, Reinkensmeyer DJ. A randomized controlled trial of gravity-supported, computer-enhanced arm exercise for individuals with severe hemiparesis. Neurorehabil Neural Repair. 2009 Jun;23(5):505-14. doi: 10.1177/1545968308331148. Epub 2009 Feb 23. PMID 19237734
- [Background] Mehrholz J, Hadrich A, Platz T, Kugler J, Pohl M. Electromechanical and robot-assisted arm training for improving generic activities of daily living, arm function, and arm muscle strength after stroke. Cochrane Database Syst Rev. 2012 Jun 13;(6):CD006876. doi: 10.1002/14651858.CD006876.pub3. PMID 22696362
- [Background] Krebs HI, Ladenheim B, Hippolyte C, Monterroso L, Mast J. Robot-assisted task-specific training in cerebral palsy. Dev Med Child Neurol. 2009 Oct;51 Suppl 4:140-5. doi: 10.1111/j.1469-8749.2009.03416.x. PMID 19740222
- [Background] Fasoli SE, Fragala-Pinkham M, Hughes R, Hogan N, Krebs HI, Stein J. Upper limb robotic therapy for children with hemiplegia. Am J Phys Med Rehabil. 2008 Nov;87(11):929-36. doi: 10.1097/PHM.0b013e31818a6aa4. PMID 18936558
- [Background] Frascarelli F, Masia L, Di Rosa G, Cappa P, Petrarca M, Castelli E, Krebs HI. The impact of robotic rehabilitation in children with acquired or congenital movement disorders. Eur J Phys Rehabil Med. 2009 Mar;45(1):135-41. PMID 19293759
- [Background] Sakzewski L, Ziviani J, Boyd R. Systematic review and meta-analysis of therapeutic management of upper-limb dysfunction in children with congenital hemiplegia. Pediatrics. 2009 Jun;123(6):e1111-22. doi: 10.1542/peds.2008-3335. Epub 2009 May 18. PMID 19451190
- [Background] Eliasson AC, Krumlinde-Sundholm L, Rosblad B, Beckung E, Arner M, Ohrvall AM, Rosenbaum P. The Manual Ability Classification System (MACS) for children with cerebral palsy: scale development and evidence of validity and reliability. Dev Med Child Neurol. 2006 Jul;48(7):549-54. doi: 10.1017/S0012162206001162. PMID 16780622
- [Background] Klingels K, De Cock P, Desloovere K, Huenaerts C, Molenaers G, Van Nuland I, Huysmans A, Feys H. Comparison of the Melbourne Assessment of Unilateral Upper Limb Function and the Quality of Upper Extremity Skills Test in hemiplegic CP. Dev Med Child Neurol. 2008 Dec;50(12):904-9. doi: 10.1111/j.1469-8749.2008.03123.x. Epub 2008 Sep 20. PMID 18811701
- [Background] Desrosiers J, Bravo G, Hebert R, Dutil E, Mercier L. Validation of the Box and Block Test as a measure of dexterity of elderly people: reliability, validity, and norms studies. Arch Phys Med Rehabil. 1994 Jul;75(7):751-5. PMID 8024419
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Gilliaux M, Lejeune T, Detrembleur C, Sapin J, Dehez B, Stoquart G. A robotic device as a sensitive quantitative tool to assess upper limb impairments in stroke patients: a preliminary prospective cohort study. J Rehabil Med. 2012 Mar;44(3):210-7. doi: 10.2340/16501977-0926. PMID 22367455
- [Background] Arnould C, Penta M, Renders A, Thonnard JL. ABILHAND-Kids: a measure of manual ability in children with cerebral palsy. Neurology. 2004 Sep 28;63(6):1045-52. doi: 10.1212/01.wnl.0000138423.77640.37. PMID 15452296
- [Background] Feldman AB, Haley SM, Coryell J. Concurrent and construct validity of the Pediatric Evaluation of Disability Inventory. Phys Ther. 1990 Oct;70(10):602-10. doi: 10.1093/ptj/70.10.602. PMID 2217539
- [Background] Noreau L, Lepage C, Boissiere L, Picard R, Fougeyrollas P, Mathieu J, Desmarais G, Nadeau L. Measuring participation in children with disabilities using the Assessment of Life Habits. Dev Med Child Neurol. 2007 Sep;49(9):666-71. doi: 10.1111/j.1469-8749.2007.00666.x. PMID 17718822